CLINICAL TRIAL: NCT05521932
Title: Establishment and Application of Endometrial 3D-organoid in Endometrial Injury Repair
Status: Completed | Type: Observational
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: Ruijin Wu
Record Dates: First submitted 2022-08-19; First posted 2022-08-30 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Asherman Syndrome
Keywords: organoid; Asherman Syndrome; intrauterine adhesion
MeSH Terms: conditions — Gynatresia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — endometrium tissue
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- IUA organoid: Organoids were generated from endometrial specimens remaining from pathological testing following adhesiolysis surgery.
  Interventions: Other: endometrium collected

INTERVENTIONS:
Other: endometrium collected — endometrium tissue collected following adhesiolysis surgery

SUMMARY:
Normal endometrial repair occurs without scar formation; however, in some women, these normal repair mechanisms are aberrant, resulting in intrauterine adhesion (IUA) formation. Intrauterine adhesion (IUA) is one of the common causes of secondary infertility, accounting for approximately 8% of disease etiologies while the pathogenesis of IUA remains unclear. Organoids derived from IUA endometrium can be used as excellent models to study IUA due to genetically stable passage and the characteristics of simulating the microenvironment of the uterine cavity.

DETAILED DESCRIPTION:
Intrauterine adhesion (IUA), also known as Asherman syndrome, is a common gynecological disease, the main clinical manifestations are oligomenorrhea, amenorrhea, recurrent miscarriage and infertility, which seriously endanger the reproductive function of women of childbearing age . Trauma and infection are the most common and important causes of IUA. At present, the incidence of infertility in the population is about 9%-18%. According to the prediction of World Health Organization (WHO), IUA will become the third largest disease after tumor and cardiovascular disease in the future.

Organoids are 3D self-organized structures that could derived from tissue and have a variety types of cell, and mimic the target organ in structure and function. They have the ability to proliferate, differentiate and self-renew. Maintain genetic stability and reproduce some physiological functions. Organoids forms closer intercellular connections and biological communication than 2D cultured cells, and is better used to simulate the occurrence process and physiological and pathological states of organs and tissues.

Therefore, investigator proposed to establish a IUA organoids bio-bank for further investigation of pathogenesis of IUA and seek for personalized therapy.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of IUA
* undergoing hysteroscopic surgery for treatment

Exclusion Criteria:

·receiving sex hormone therapy in the three months before surgery

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients undergoing intrauterine adhesiolysis surgery at the Department of Gynecology of the Women's Hospital, School of Medicine, Zhejiang University
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
IUA organoid formation efficiency | 2 years
  Establishment IUA organoid from patient-derived endometrium tissue. The following outcome measure would be calculated:
  * the formation efficiency of organoid
IUA organoid proliferative rate | 2 years
  Establishment IUA organoid from patient-derived endometrium tissue. The following outcome measure would be calculated:
  * the proliferative rate of organoid

SECONDARY OUTCOMES:
IUA organoid identification | 2 years
  the IUA organoid identification will assessed by the following method: Identification of cell type and ultrastructure of IUA organoid by pathological staining and electron microscope.

CONTACTS AND LOCATIONS:
Overall Officials: Ruijin Wu, M.D., Study Chair — Women's Hospital, College of Medicine Zhejiang University
Locations (1):
- Women's Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided